CLINICAL TRIAL: NCT01891162
Title: Socioeconomic Profile and QUALITY OF LIFE FOR WOMEN WITH AND WITHOUT PELVIC FLOOR DYSFUNCTION
Brief Title: Assessment of Socioeconomic Status by Brazil and Quality of Life for Urinary Incontinence in Brazilian Women
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ISADRI
Record Dates: First submitted 2013-03-08; First posted 2013-07-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Incontinence Urinary
Keywords: quality of life, incontinence urinary, socioeconomic
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Assessment will be carried out general quality of life beyond the functional evaluation of the pelvic floor through the PERFECT
- Study: Will be held evaluate the quality of life for general and specific pelvic floor dysfunction beyond the functional assessment of the pelvic floor through the PERFECT.

SUMMARY:
Age, parity, obesity and a number of comorbidities are the major clinical and lifestyle risk factors for female urinary incontinence and pelvic organ prolapse at the population level. The socioeconomic risks for incontinence have however, conflicting evidence with assorted measures of socioeconomic status. Brazil is a country with enormous social contrasts, and deep inequality. We have a mixed origin of cultures and different economic and regional conditions. We believe that the perception and the impact that has Pelvic floor dysfunction in the quality of life of the woman must vary widely according to socioeconomic status (including household income, highest educational level, family income). There is to date no studies have correlated a criterion for classifying economic official in Brazil with the impact of quality of life (based in KHQ or PQOL) of women with urinary incontinence and pelvic organ prolapse.

DETAILED DESCRIPTION:
The research is being conducted at the Department of Gynecology of a referral hospital in the state of Ceará, Brazil in the period October 2011 to February 2012. Women will be referred from Primary Care and Health scheduled for evaluation in the sector of Urogynecology Cesar Cals General Hospital, Department of Health of the State of Ceará. During the study period 200 patients will be treated with complaints of urinary incontinence or pelvic organ prolapse in the sector. Included in the study women who were postmenopausal, who are not taking hormone therapy in the last six months. Women with urinary loss, which does not have non-inhibited contraction of the detrusor proven by urodynamic study. Will be compared with a group of women without pelvic floor dysfunction confirmed by clinical history and gynecological examination with the same characteristics in relation to postmenopausal status, all from the general gynecology outpatient clinic. Will be used for data collection socioeconomics an interview administrated questionnaire adapted from the Brazil Economic Classification Criterion - 2011 (CCEB) The CCEB is an instrument of economic segmentation that uses the survey of household characteristics (presence and quantity of some items of comfort and home schooling level of household head) to differentiate the population. The criterion assigns points according to each household characteristic and performs the sum of these points. Then will be made a match score of the test strips and layers of economic status defined by A1, A2, B1, B2, C1, C2, D, E. This criterion was designed to define broad classes that meet the needs of segmentation (by purchasing power) of most companies. To evaluate Quality of Life in Urinary incontinence and pelvic organ prolapse women we used the KHQ questionnaire, QoL-P respectively. To evaluate the Overall Quality of Life, SF-36. For functional evaluation of the pelvic floor (AP) bidigital evaluation was performed using the classification of Ortiz (1996) and schema PERFECT Oxford (1990). Will be used the application EpiInfo version 6.04, Atlanta, USA. Will be studied the socioeconomic variables (age, educational level, economic status and income), health perception variables (the impact of incontinence / prolapse, the limitations of performance tasks, physical limitation, social limitation, personal relationships, the emotions, sleep and energy and gravity measurements). Will be used the prevalence of urinary incontinence as a measure of the occurrence and chi-square test and test of Pearson to evaluate the statistical significance considering p <0.05. Exploratory analysis will also performed to describe the frequency distribution of socioeconomic variables.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* clinical diagnosis of urinary incontinence and / or pelvic organ prolapse
* without contraction uninhibited detrusor

Exclusion Criteria:

* cognitive deficit
* presence of uninhibited detrusor contraction

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: will be avalueted women who will be postmenopausal, who are not taking hormone therapy in the last six months. Women with urinary loss, which does not have non-inhibited contraction of the detrusor proven by urodynamic study. Will be compared with a group of women without pelvic floor dysfunction confirmed by clinical history and gynecological examination with the same characteristics in relation to postmenopausal status, all from the general gynecology outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of socioeconomic status by Brazil and quality of life for urinary in Brazilian women | one year

CONTACTS AND LOCATIONS:
Overall Officials: ISABELLA P FROTA, Principal Investigator — Pesquisadora
Locations (2):
- Brazil (2):
  - Cesar cals hospital, Fortaleza, Ceará
  - General Hospital Fortaleza, Fortaleza, Ceará